CLINICAL TRIAL: NCT04907292
Title: Quality of Recovery After Unplanned and Planned Cesarean Deliveries - an Application of ObsQoR-10
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21-04
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2021-09

CONDITIONS: Quality of Recovery
Keywords: Cesarean delivery; ObsQoR-10©

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Planned Cesarean delivery: Patients who have an elective Cesarean delivery at Mount Sinai Hospital
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool
- Unplanned Cesarean delivery: Patients who have an unplanned Cesarean delivery at Mount Sinai Hospital
  Interventions: Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool

INTERVENTIONS:
Other: Obstetric Quality of Recovery-10 (ObsQoR-10©) Scoring Tool — The ObsQoR-10 tool aims to quantitatively measure functional recovery at 24 hours postpartum. It includes 10 questions on a 0 to 10 scale, aimed at pain management, the adverse effects of narcotics and the perception of recovery by the patient.
  Other Names: ObsQoR-10©

SUMMARY:
In Canada, 29.1% of annual births are via cesarean deliveries (CD). The literature shows that almost 24% of CDs are unplanned. Existing evidence suggests that unplanned cesarean delivery, compared to elective cesarean, may be associated with poor maternal recovery, longer postpartum hospital stays and more opioid requirements after surgery. Since the establishment of the Enhanced Recovery After Cesarean protocols, specific care pathways have been implemented with the aim of optimizing recovery after CD and to reduce the costs to the health care system. However, the majority of unplanned cesarean receive the same postoperative anesthetic, obstetric and nursing care as the elective CDs.

Looking at the actual information about maternal recovery after unplanned CD, the investigators found that there is a paucity of literature examining this topic utilizing validated, patient-oriented quality of recovery tools. Recently, Obstetric Quality of Recovery-10 scoring tool (ObsQoR-10), a new patient-focused outcome instrument for postpartum recovery, it has been validated for all types of deliveries, in the inpatient setting. ObsQoR-10 tool aims to measure quantitatively functional recovery at 24 hours postpartum. It includes 10 questions on a 0 to 10 scale, aimed at pain management, the adverse effects of narcotics and the perception of recovery by the patient.

The aim of this study is to determine the quality of recovery from unplanned cesarean deliveries compared to planned ones using a validated tool for recovery after cesarean delivery (ObsQoR-10 tool).

The investigators hypothesize that quality of recovery as measured by the Obs-QoR10 for unplanned cesarean deliveries will be lower than the planned CDs.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years old and over
* Term singleton pregnancy
* Undergoing planned or unplanned caesarean delivery at Mount Sinai Hospital
* Patients who have given informed written consent

Exclusion Criteria:

* Patients who have refused, are unable to give or have withdrawn consent
* Patients unable to communicate fluently in English
* Patients with American Society of Anesthesiologists (ASA) classification of 4 or greater
* Patients scheduled to have a classical vertical incision
* Patients undergoing cesarean hysterectomy
* Patients with history of chronic pain, chronic use of analgesic drugs, or history of opioid or intravenous drug abuse
* Patients who have refused neuraxial anesthesia, or those in whom it is contraindicated.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who deliver by planned or unplanned cesarean section at Mount Sinai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-09 (Actual)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) score 24 hours | 24 hours
  ObsQoR-10 score at 24 hours after surgery for both planned and unplanned cesarean deliveries. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.

SECONDARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) score 48 hours | 48 hours
  ObsQoR-10 score at 48 hours after surgery for both planned and unplanned cesarean deliveries. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.
Obstetric Quality of Recovery-10 (ObsQoR-10) score 7 days | 7 days
  ObsQoR-10 score at 7 days after surgery for both planned and unplanned cesarean deliveries. There are 10 questions, and the results are tabulated out of 100. The higher the overall score out of 100, the better quality of recovery a patient is experiencing.
Pain Score (VAS) - 24 hours | 24 hours
  Verbal analogue scale (VAS) of 0-10, where 0= no pain and 10=worst pain imaginable, at 24 hours post cesarean delivery
Pain Score (VAS) - 48 hours | 48 hours
  Verbal analogue scale (VAS) of 0-10, where 0= no pain and 10=worst pain imaginable, at 48 hours post cesarean delivery
Opioid consumption - 24 hours | 24 hours
  Total opioid consumption within 24 hours post cesarean
Opioid consumption - 48 hours | 48 hours
  Total opioid consumption within 48 hours post cesarean
Hospital discharge - questionnaire, 24 hours | 24 hours
  At 24 hours post cesarean, patients will be asked the question "Are you ready to be discharged from the hospital? Yes or No"
Hospital discharge - questionnaire, 48 hours | 48 hours
  At 48 hours post cesarean, patients will be asked the question "Are you ready to be discharged from the hospital? Yes or No"

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No